CLINICAL TRIAL: NCT03452709
Title: Clinical Trial of the Effectiveness of Non-pharmacological Interventions (Physical Activity + ABPM) in Patients With Cardiovascular Risk Factors in Primary Care
Brief Title: Effectiveness of Non-pharmacological Interventions in Patients With Cardiovascular Risk Factors in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: MurciaSalud (Other Government); Public Health Service, Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTIVA
Record Dates: First submitted 2011-06-22; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2017-12

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease;; primary prevention;; physical activity;; Blood Pressure Monitoring, Ambulatory
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group: no intervention (No Intervention): Only the normal practise
- therapeutic exercise (Experimental): In this group the intervention is the prescription of physical activity. The duration of the groups is planned to be from 12 weeks with 3 programmed sessions per week.
  Interventions: Behavioral: therapeutic exercise
- ABPM (Experimental): In this group the arterial pressure is evaluated with ABPM.
  Interventions: Device: ABPM ambulatory blood pressure monitoring
- therapeutic exercise + ABPM (Experimental)
  Interventions: Behavioral: therapeutic exercise; Device: ABPM ambulatory blood pressure monitoring

INTERVENTIONS:
Behavioral: therapeutic exercise — The duration of the groups is planned to be from 12 weeks with 3 programmed sessions per week. physical activity programmed by an instructor in patient with high risk of cardiovascular.
  Arms: therapeutic exercise; therapeutic exercise + ABPM
Device: ABPM ambulatory blood pressure monitoring — Arterial pressure is a biological variable which fluctuates over a 24 hour period depending on the period of activity/rest, which is known as circadian the BP rhythm. Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) vary, on average, more than 50 mm Hg throughout the day in a normotensive adult.
  Arms: ABPM; therapeutic exercise + ABPM

SUMMARY:
The principal objective is analyzed whether a selective intervention no pharmacological (use of ABPM +/- prescription of physical exercise) for cardiovascular risk factors in patients with high cardiovascular risk in primary prevention is associated with a decrease in cardiovascular risk measured using the risk Score tables for countries with a low risk. It will be independently analized the effectiveness of systematic use of ABPM and the prescription of physical exercise.

DETAILED DESCRIPTION:
Cardiovascular disease continues to be the main cause of death in Western countries, with a very high prevalence (affecting >1 in every 3 adult Americans), and contributes as one of the highest annual healthcare costs. There is still enormous potential for improving prevention although notable efforts have already been made. In the Spanish population, the following cardiovascular risk factors have been identified as being most prevalent: arterial hypertension, dyslipidemia, having a sedentary lifestyle, tobaccoism, obesity and diabetes.

Essential Arterial Hypertension (EAH) is the most prevalent cardiovascular risk factor in the world and the main cause of cardiovascular disease. There are many clinical practice guides which recommend carrying out moderate physical activity to prevent, delay or reduce hypertension, given that the practice of community interventions with physical activity have been efficient.

The indication to perform Itinerant Monitorization blood pressure in the diagnosis of hypertension is included in the latest draft of the clinical practice guideline from NICE, National Institute for Health and Clinical Excellence .

Other cardiovascular risk factor to take into account is dyslipidemia, the prevalence of dyslipidemia is 16.2% in adults aged over 20 years. For this condition, physical activity is also recommended.

When faced with a sedentary lifestyle or physical inactivity two intervention measures are available for reducing its incidence: verbal healthcare advice (taking advantage of the patients visit to the consultation) and the prescription of physical exercise.

Taking into account the interventions mentioned that can be carried out in the face of risk factors, and that a multifactorial intervention is more efficient that individual interventions, the investigators have designed a clinical trial which attempts to improve most of the principal risk factors. The objective is to reduce the cardiovascular risk of patients using a multifactorial intervention on hypertension, dyslipidemia, sedentary lifestyle. The investigators will evaluate the efficiency of a program for official prescriptions for physical exercise compared to structured verbal advice in hypertense patients undergoing treatment and who have another risk factors (dyslipidemia being treated for more than one year or they are smokers), including action to improve the treatment adaptation for the hypertension (ABPM).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing treatment with at least one hypertense drug due to HTA and at least one hypolipemiant drug prescribed due to hypercholesterolemia, or other risk factor. The treatment should have a minimum duration time of 12 months prior to inclusion in the study.
* Patient in Primary Prevention.
* Finding oneself in the sedentary lifestyle category or through activation of the simplified active questionnaire of physical activity extracted from the Lipid Research Clinics prevalence Study

Exclusion Criteria:

* Serious or terminal diseases.
* Diagnosis of ischemic and/or cerebrovascular cardiopathy.
* Patients with a limiting pathology which prevents physical exercise being performed.
* Serious mental illnesses: Psychosis, Major depressive disorder, Neurosis.
* Diabetes mellitus.
* Patients with limiting pathology preventing them from carrying out physical exercise.
* Serious mental diseases: Psychosis, Major depresive disorder, Neurosis.
* Pregnancy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3656 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk . | Every 3 months , up to 12 months.
  Tables for countries with low cardiovascular risk
Systolic arterial tension | Every 3 months , up to 12 months
  blood pressure

SECONDARY OUTCOMES:
diastolic arterial tension | Every 3 months , up to 12 months
  blood pressure
Cholesterol levels. | Every 3 months , up to 12 months
  blood levels.
Physical Activity | Every 3 months , up to 12 months
  International Physical Activity Questionniare (IPAQ) 600-3000 MET (METs are multiples of the resting metabolic rate
Pharmacological treatment. | Every 3 months , up to 12 months
  Number of antihypertensive and hypolipemiant drug and dose.
EUROFIT battery | Every 3 months , up to 12 months
  Score obtained

CONTACTS AND LOCATIONS:
Overall Officials: A LOPEZ-SANTIAGO, MD, Principal Investigator — Consejeria de sanidad y consumo, Direccion general de planificacion, ordenacion sanitaria y farmaceutica e investigacion.
Locations (1):
- Fundación para la Formación e Investigación Sanitarias de la Región de Murcia, Murcia, Murcia, Spain

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Medrano MJ, Cerrato E, Boix R, Delgado-Rodriguez M. [Cardiovascular risk factors in Spanish population: metaanalysis of cross-sectional studies]. Med Clin (Barc). 2005 Apr 30;124(16):606-12. doi: 10.1157/13074389. Spanish. PMID 15871776
- [Background] Stamler J, Vaccaro O, Neaton JD, Wentworth D. Diabetes, other risk factors, and 12-yr cardiovascular mortality for men screened in the Multiple Risk Factor Intervention Trial. Diabetes Care. 1993 Feb;16(2):434-44. doi: 10.2337/diacare.16.2.434. PMID 8432214
- [Background] Ezzati M, Lopez AD, Rodgers A, Vander Hoorn S, Murray CJ; Comparative Risk Assessment Collaborating Group. Selected major risk factors and global and regional burden of disease. Lancet. 2002 Nov 2;360(9343):1347-60. doi: 10.1016/S0140-6736(02)11403-6. PMID 12423980
- [Background] Martin-Baranera M, Campo C, Coca A, de la Figuera M, Marin R, Ruilope LM; en representacion del Grupo de Investigadores DICOPRESS. [Stratification and degree of control of cardiovascular risk factors in hypertensive Spanish population. Results of the DICOPRESS study]. Med Clin (Barc). 2007 Jul 14;129(7):247-51. doi: 10.1157/13108347. Spanish. PMID 17683705
- [Background] Sierra C, De la Sierra A, Sobrino J, Segura J, Banegas JR, Gorostidi M, Ruilope LM; en representacion de los Investigadores del Registro Nacional de MAPA. Sociedad Espanola de Hipertension-Liga Espanola para la Lucha contra la Hipertension Arterial (SEH-LELHA). [Ambulatory blood pressure monitoring (CABPM): clinical characteristics of 31,530 patients]. Med Clin (Barc). 2007 Jun 2;129(1):1-5. doi: 10.1157/13106673. Spanish. PMID 17570178
- [Background] Hypertension: clinical management of primary hypertension in adults NICE guideline. Draft for consultation, February 2011. access (29/3/2011: http://www.nice.org.uk/nicemedia/live/12167/53225/53225.pdf).
- [Background] Lee LL, Arthur A, Avis M. Evaluating a community-based walking intervention for hypertensive older people in Taiwan: a randomized controlled trial. Prev Med. 2007 Feb;44(2):160-6. doi: 10.1016/j.ypmed.2006.09.001. Epub 2006 Oct 20. PMID 17055561
- [Background] Elley CR, Garrett S, Rose SB, O'Dea D, Lawton BA, Moyes SA, Dowell AC. Cost-effectiveness of exercise on prescription with telephone support among women in general practice over 2 years. Br J Sports Med. 2011 Dec;45(15):1223-9. doi: 10.1136/bjsm.2010.072439. Epub 2010 Nov 16. PMID 21081641
- [Background] Grandes G, Sanchez A, Sanchez-Pinilla RO, Torcal J, Montoya I, Lizarraga K, Serra J; PEPAF Group. Effectiveness of physical activity advice and prescription by physicians in routine primary care: a cluster randomized trial. Arch Intern Med. 2009 Apr 13;169(7):694-701. doi: 10.1001/archinternmed.2009.23. PMID 19364999
- [Background] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh/68002318
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh?term=PRIMARY%20PREVENTION
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh?term=physical%20activity
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh/68018660